CLINICAL TRIAL: NCT04791241
Title: Evaluation of a Check-list Including Lung Ultrasound for the Management of Patients With Acute Respiratory Failure at the Emergency Department During the COVID-19 Era
Brief Title: A Check-list Including Lung Ultrasound for ED Patients With ARF
Acronym: CHECKIRA-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHMS20005
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Failure
Keywords: Covid19; Acute Respiratory Failure; Ultrasound; Checklist; Emergency; Diagnosis
MeSH Terms: conditions — COVID-19; Emergencies; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- check-list with ultrasound (Experimental): check-list including lung ultrasound for the management of patients with acute respiratory failure at the emergency department during the COVID-19 era
  Interventions: Other: check-list including lung ultrasound

INTERVENTIONS:
Other: check-list including lung ultrasound — The investigator will follow the checklist which includes the collection of anamnestic data and clinical signs, the performance of a pulmonary embolism clinical probability score and a cardiopulmonary ultrasound with count -standardized rendering. After completing this checklist, the investigator will note their diagnosis (list of proposals on the data collection sheet), the treatments started (closed list of therapeutic classes). If he orders other tests, he will write them down and then note the diagnosis made and the treatments prescribed after obtaining the results of these tests.
  The therapeutic management of patients compared to the usual care in the respective departments may be modified depending on the results of the cardiopulmonary ultrasound . The emergency physician may initiate therapy before the results of additional examinations that he would have usually performed without cardiopulmonary ultrasound.

SUMMARY:
The aim of the study is to evaluate if a check-list including lung ultrasonography can help to identify the etiology of the acute respiratory failure of patients managed at the emergency room.

Adult patients admitted to the emergency room for acute respiratory failure will be offered the study. The emergency physician will perform a systematic examination using a checklist, including pulmonary embolism prediction scores, structured clinical examination and lung ultrasound, in order to establish a diagnostic hypothesis.

A diagnostic hypothesis will be made after completion of the checklist. The emergency physician can perform additional examinations and treatment after completion of the checklist.

The final diagnosis will be checked by an adjudication committee which will have all the documents established during the emergency room consultation and any hospitalization following this hospitalization.

The main outcome will be the concordance rate between the diagnosis after the check-list and the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute respiratory failure table (SpO2 90% in ambient air or need more than 3 L/min of oxygen to have SpO2 > 92% AND/OR signs of respiratory struggle sign AND/OR respiratory rate control > 25 cycles/minute AND/OR cyanosis)
* Over 18 years old

Exclusion Criteria:

* Pregnant, Parturising or Breastfeeding Women
* Patient who has already participated in the study in the previous 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Agreement between the etiology retained after using the checklist and the diagnosis retained by an adjudication committee after analysis of the entire patient file. | 1 month after inclusion
  The adjudication committee will meet all 35 inclusions to determine the diagnosis of each patient after analysis of the complete anonymized file which will be provided by locol investigator one month after inclusion.

SECONDARY OUTCOMES:
Analysis of the diagnosis retained after the checklist in patients with a final diagnosis of COVID-19; analysis of the final diagnosis in patients with a diagnosis of COVID-19 evoked after the checklist | One month after inclusion
  The adjudication committee will meet periodically after analysis of the complete anonymized file to check the COVID diagnosis.
Collection of treatments started only after completion of the checklist and verification of its suitability for the diagnosis selected | at one day
  All the treatments started only after completion of the checklist wil be collected prospectively and their appropriateness will be checked.
Collection of additional examinations possibly performed in the emergency unit after the completion of the checklist | at one day
  All additional examinations performed after the completion of the checklist will be collected
Comparison of treatments introduced after completion of the checklist and after the other additional examinations performed at the emergency room | at one day
  all treatments delivered after the completion of the checklist and after complementary exams will be collected and classified into therapeutic families (antibiotics, diuretics).
Delay between completion of the checklist and obtaining the results of any other examinations | At one day
  Time between the completion of the checklist and obtaining the last result of the other examinations performed at the emergency room (except for bacterial culture)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Annecy Genevois, Annecy
  - Centre Hospitalier Metropole Savoie, Chambéry
  - CHUGA, Grenoble

IPD SHARING:
Plan to Share IPD: No